CLINICAL TRIAL: NCT01873612
Title: Acute Ventilatory Response to Hypoxia During Sedation With Dexmedetomidine Compared to Propofol in Healthy Male Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PropDexHVRVolunteers
Record Dates: First submitted 2013-05-29; First posted 2013-06-10 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Hypoxia; Anesthetics; Conscious Sedation; Hypercapnia
Keywords: Dexmedetomidine; Propofol; Hypoxic ventilatory response; Hypercapnic ventilatory response
MeSH Terms: conditions — Hypoxia; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedation with dexmedetomidine (Experimental): Sedation with dexmedetomidine
  Interventions: Procedure: Hypoxic ventilatory response; Procedure: Hypercapnic ventilatory response
- Sedation with propofol (Experimental): Sedation with propofol
  Interventions: Procedure: Hypoxic ventilatory response; Procedure: Hypercapnic ventilatory response

INTERVENTIONS:
Procedure: Hypoxic ventilatory response
  Other Names: HVR
Procedure: Hypercapnic ventilatory response
  Other Names: HCVR

SUMMARY:
The overall aim with this project is to investigate the effect of dexmedetomidine on control of breathing in healthy volunteers and to compare it with propofol at the same degree of sedation.

DETAILED DESCRIPTION:
15 volunteers will be investigated for their hypoxic and hypercapnic ventilatory response during sedation with dexmedetomidine and propofol in a randomized cross-over study.

6 volunteers will be investigated for their repeated response to hypoxia and hypercapnia in order to validate the method.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 18-40
3. American Society of Anesthesiologist´s classification (ASA) 1, i.e. healthy
4. No medication
5. No allergies
6. Non-smoker/no snuff, i.e. no nicotine intake
7. Normal weight, BMI <26

Exclusion Criteria:

Snoring

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Hypoxic ventilatory response | One day for each drug; before,during and after sedation with dexmeditomidine or propofol
  Acute hypoxic ventilatory response,i.e. the ventilatory response to acute hypoxia measured as change in minute ventilation over change in peripheral oxygen saturation

SECONDARY OUTCOMES:
hypercapnic ventilatory response | One day for each drug; Before, during and after sedation with dexmedetomidine or propofol
  The acute ventilatory response to hypercapnia, i.e. change in minute ventilation over change in end-tidal carbon dioxide

OTHER OUTCOMES:
upper airway obstruction | One day for each drug: Before, during and after sedation with dexmedetomidine or propofol
  Objective signs of upper airway obstruction, e.g. Interruption of airflow at the same time as breathing movements of the thoracic wall, paradoxal breathing, increased airway resistance
Plasma concentration | One day for each drug; At target sedation
  Plasma concentration of dexmedetomidine or propofol
Sedation level | One day; During the whole experimental procedure
  Sedation level will be measured as Richmond Agitation Sedation Scale(RASS) the observer's assessment of alertness/sedation scale (OAA/S)
Bispectral index | One day; During the whole experimental procedure
  Bispectral index (BIS) gives a number between 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, MD, PhD, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Department of Anesthesiology, Surgical Sciences and Intensive Care Medicine, Karolinska University Hospital, Stockholm, Sweden